CLINICAL TRIAL: NCT03855345
Title: Antimicrobial Photodynamic Therapy Mediated by PapaMBlue® on Chronic Periodontal Disease - Randomized Blind Controlled Trial
Brief Title: Antimicrobial Photodynamic Therapy Mediated by PapaMBlue® on Chronic Periodontal Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Renato Araujo Prates, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIU
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be present during the treatments, so he will not know to which group the participants belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): In this group, the participants will be submitted to the conventional treatment. The treatment will consist of oral hygiene orientation, with instructions of brushing technique and recommendation of the daily use of dental floss. All patients will receive a demonstration of oral hygiene techniques. The calculus deposits on the teeth will be removed with ultrasound equipment and curettes for root scaling and straightening. After the use of ultrasound and curettes, bicarbonate jet will be used to remove dental biofilm. Treatment will be performed in 2 to 4 sessions under local anesthesia (typically 2% mepivacaine with 1: 100,000 noradrenaline). Gracey periodontal curettes (numbers 3/4, 7/8, 11/12 and 13/14) and Mc Call curettes for removal of the dental calculus will be used. Other biofilm-retaining factors, such as carious lesions, condemned teeth, and ill-adapted restorations, will be removed during these periodontal treatment sessions.
  Interventions: Procedure: Conventional treatment
- aPDT group (Experimental): In this group, besides the conventional treatments, patients will also receive aPDT. aPDT will be performed at the end of each periodontal treatment session, at sites with bags greater than or equal to 4 mm. The photosensitizer PapaMBlue® (F & A Ltda, São Paulo, Brazil) will be deposited in the pouches with a syringe, with the application in coronal direction, and a time of 1 min of pre-irradiation will be adopted so that the substance can stain bacterial biofilm (according to the manufacturer's information). Next, the diode laser emitting wavelength of ʎ=660 nm, with power of P=100 mW, will be applied. The laser will be applied to the mucosa, over the oral epithelium with an optical fiber. Irradiation will be performed until the entire periodontal pocket is illuminated for 2 min at each point. Each irradiation point will be approximately 0.4cm2, which will result in energy density of 30 J/cm2 in 2 min irradiation. The irradiation will have a constant power density of 250 mW/cm2.
  Interventions: Procedure: Conventional treatment; Radiation: aPDT

INTERVENTIONS:
Procedure: Conventional treatment — The treatment will consist of oral hygiene orientation, with instructions of brushing technique and recommendation of the daily use of dental floss. All patients will receive a demonstration of oral hygiene techniques. The calculus deposits on the teeth will be removed with ultrasound equipment and curettes for root scaling and straightening. After the use of ultrasound and curettes, bicarbonate jet will be used to remove dental biofilm. Treatment will be performed in 2 to 4 sessions under local anesthesia (typically 2% mepivacaine with 1: 100,000 noradrenaline). Gracey periodontal curettes (numbers 3/4, 7/8, 11/12 and 13/14) and Mc Call curettes for removal of the dental calculus will be used. Other biofilm-retaining factors, such as carious lesions, condemned teeth, and ill-adapted restorations, will be removed during these periodontal treatment sessions.
Radiation: aPDT — aPDT will be performed at the end of each periodontal treatment session, at sites with bags greater than or equal to 4 mm. The photosensitizer PapaMBlue® (F & A Ltda, São Paulo, Brazil) will be deposited in the pouches with a syringe, with the application in coronal direction, and a time of 1 min of pre-irradiation will be adopted so that the substance can stain bacterial biofilm (according to the manufacturer's information). Next, the diode laser emitting wavelength of ʎ=660 nm, with power of P=100 mW, will be applied. The laser will be applied to the mucosa, over the oral epithelium with an optical fiber. Irradiation will be performed until the entire periodontal pocket is illuminated for 2 min at each point. Each irradiation point will be approximately 0.4cm2, which will result in energy density of 30 J/cm2 in 2 min irradiation. The irradiation will have a constant power density of 250 mW/cm2.
  Arms: aPDT group

SUMMARY:
The elimination of the pathogenic microorganisms of the periodontal pocket is one of the main points for success in periodontal treatment. The objective of this study is to investigate the clinical and antimicrobial effect of papain-mediated photodynamic therapy in the clinical treatment of periodontal disease. Twenty patients with chronic periodontitis will be selected. Patients will be divided randomly into two groups (n = 10), and the control group will receive conventional periodontal treatment and group II will receive conventional treatment and antimicrobial photodynamic therapy (aPDT). Conventional treatment will consist of oral hygiene guidance, with brushing technique instructions and recommendation of daily flossing. The calculus deposits on the teeth will be removed with ultrasound equipment and curettes for scraping and root planing. The aPDT will be performed at the end of each periodontal treatment session, at sites with bags greater than or equal to 4 mm. The PapaMblue® photosensitizer will be deposited in the periodontal pockets with a syringe and a pre-irradiation time of 1 min will be adopted. Then, the laser emitting wavelength of 660 nm, with power of 100 mW, for 2 min, radiant exposure of 30 J/cm2 and power density of 250 mW/cm2 will be applied. Patients will undergo clinical evaluations before treatment (day 1) and 30, 60 and 90 days after the end of treatment. Microbiological evaluations will be made before and 30 days after treatment. The distribution of the data within each group and the homogeneity of the variances will be verified. With this information, the most appropriate statistical test for each evaluation will be used. The sample calculation is based on the literature and the significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have chronic periodontitis (AAP, 2001);
* At least 10 present teeth, with at least 3 sites with clinical depth of probing greater than 4 mm;
* The patient must be in periodontal treatment at the Dental Clinic of Universidade Nove de Julho, institution where this research will be carried out;

Exclusion Criteria:

* Smokers or former smokers who discontinued the habit less than 12 months prior to selection;
* Uncontrolled diabetes;
* Anemia;
* Cancer;
* Pregnant women;
* Use of antibiotics in the last 6 months;
* Use of anti-inflammatory in the last 3 months;
* Coagulation disorder (use of anti-coagulant, presence of liver diseases, thrombocytopenia and immunosuppression);
* Patients under orthodontic treatment;
* Patients who maintain a biofilm index greater than 25%.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in probing depth | Baseline, 30, 60 and 90 days after treatment.
  For the evaluation of probing depth, a single trained, calibrated examiner will examine 6 sites of each tooth with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of probing depth in milimeters. The evaluation will be performed at the beginning of treatment, 30, 60 and 90 days after the tretaments.

SECONDARY OUTCOMES:
Change in probing bleeding | Baseline, 30, 60 and 90 days after treatment.
  For the evaluation of bleeding, a single trained, calibrated examiner will examine 6 sites of each tooth using a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) to check whether there is bleeding during the probing. The evaluation will be performed at the beginning of treatment, 30, 60 and 90 days after the treatments.
Change in loss of clinical insertion | Baseline, 30, 60 and 90 days after treatment.
  A single trained, calibrated examiner will examine 6 sites in each tooth with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of loss of clinical insertion in milimeters. The evaluation will be performed at the beginning of treatment, 30, 60 and 90 days after the treatments.
Change in plaque index | Baseline, 30, 60 and 90 days after treatment.
  For the evaluation of plaque index, a single trained, calibrated examiner will examine 6 sites of each tooth with a 15mm North Carolina millimeter probe (Hu-Friedy, Chicago, IL, USA) for the measurement of the amount of plaque in milimeters. The evaluation will be performed at the beginning of treatment, 30, 60 and 90 days after treatment.
Microbiological examination (change in CFUs (Colony Forming Units)) | Baseline, 30, 60 and 90 days after treatment.
  The microbiological examination will be performed from subgingival biofilm samples collected from the periodontal pockets. Two collections will be performed at each experimental site before and immediately after treatments. For the collection of the subgingival biofilm, a relative isolation of the teeth with cotton rollers will be performed, the supra-gingival biofilm will be removed with sterile gauze, and the subgingival biofilm sample will be obtained by inserting a sterile absorbent paper tip (no. 30) into the inside of the pocket, being held in place for 30s. The tips will be removed and stored in properly identified sterile plastic microtubes, with each paper cone being stored in a different microtube.
  The samples will be used to determine the CFUs (Colony Forming Units).